CLINICAL TRIAL: NCT05023629
Title: STunning After Balloon Occlusion, A Single-center, Single-arm, Prospective Study
Brief Title: STunning After Balloon Occlusion
Acronym: STABO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: v.2.0
Record Dates: First submitted 2021-07-05; First posted 2021-08-26 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous Coronary Intervention; Myocardial stunning
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Stunning

STUDY DESIGN:
Intervention Model Description: A single-center, single-arm, prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with a significant coronary artery lesion (Other): Balloon inflation for 90s
  Interventions: Other: Intracoronary balloon inflation

INTERVENTIONS:
Other: Intracoronary balloon inflation — Patients with a significant coronary artery lesion in a proximal coronary segment will undergo intracoronary balloon inflation for 90s prior to PCI.

SUMMARY:
The aim of this study is to examine in-depth cardiac function and morphology after short-term coronary occlusion by balloon inflation in patients with stable coronary artery disease (CAD) who undergo percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
Primary objectives:

1. To determine the time-course for the resolution of regional myocardial function after short-term coronary artery occlusion in patients with stable CAD who undergo PCI.

   Secondary objectives:
2. To confirm by cardiac magnetic resonance imaging that no myocardial injury occurs after short-term coronary occlusion in patients who undergo PCI due to stable CAD.
3. To establish a clinical model for studying myocardial stunning.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years.
2. Stable CAD with indication for PCI of a lesion in either of the following coronary segments:

   1. 6 or 7 (proximal or mid left anterior descending coronary artery)
   2. 11 (Proximal left circumflex coronary artery)
   3. 1 or 2 (proximal right coronary artery)
3. Normal cardiac function in the myocardial segments subtended by the target vessel, as assessed by echocardiography at the time of coronary angiography.
4. Written informed consent obtained.

Exclusion Criteria:

1. Pre-existing heart failure
2. Known pre-existing irreversible regional or global wall motion abnormalities affecting the myocardial segments subtended by the target vessel.
3. Severe valvulopathy
4. Thrombolysis In Myocardial Infarction (TIMI) flow <3 in the target vessel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Precent Akinesia | 30 minutes post balloon occlusion
  Time until recovery of percent akinesia (percent Akinesia; defined as more than 80 percent recovery compared to percent Akinesia at 30 minutes post balloon occlusion).

SECONDARY OUTCOMES:
Difference in percent Akinesia | 30 minutes
  Difference in percent Akinesia at 30 minutes compared to baseline (before balloon occlusion).
Difference in radial myocardial Strain | 30 minutes
  Difference in radial myocardial Strain (in percent) in the myocardial segments subtended by the target vessel at 30 minutes compared to baseline measured with speckle tracking.
Time until recovery of radial Strain | 30 minutes
  Time until recovery of radial Strain in the myocardial segments subtended by the target vessel (defined more than 80 percent recovery compared to 30 minutes post balloon occlusion)
Percent Akinesia | 1, 10, 30, 60, 120, 180 and 300 minutes and 24, 48 and 72 hours
  Percent Akinesia in the myocardial segments
Radial myocardial Strain | 1, 10, 30, 60, 120, 180 and 300 minutes and 24, 48 and 72 hours
  Radial myocardial Strain (in percent) in the myocardial segments subtended by the target vessel measured with speckle tracking.
Global longitudinal Strain | 1, 10, 30, 60, 120, 180 and 300 minutes and 24, 48 and 72 hours
  Global longitudinal Strain (in percent) in the heart measured with speckle tracking.
Myocardial wall motion index | 1, 10, 30, 60, 120, 180 and 300 minutes and 24, 48 and 72 hours
  Myocardial wall motion index
Left ventricular ejection fraction | 1, 10, 30, 60, 120, 180 and 300 minutes and 24, 48 and 72 hours
  Left ventricular ejection fraction
Left ventricular stroke volume index | 1, 10, 30, 60, 120, 180 and 300 minutes and 24, 48 and 72 hours
  Left ventricular stroke volume index

CONTACTS AND LOCATIONS:
Overall Officials: Björn Redfors, Principal Investigator — Sahlgrenska Universitetssjukhus
Locations (1):
- Kardiologen, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No
Due to GDPR regulation